CLINICAL TRIAL: NCT03019679
Title: Serum Endocan Levels in Polycystic Ovary Syndrome: a Possible Marker of Angiogenic Dysfunction
Brief Title: Serum Endocan Levels in Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, İlhan Bahri Delibas, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: GaziosmanpasaU
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — serum samples,centrifuged
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study group: Patients with polycystic ovary syndrome
- Control group: Patients without polycyctic ovary syndrome

SUMMARY:
In this study the investigators aimed to investigate whether there is a relation between polycystic ovary syndrome and serum endocan levels.

DETAILED DESCRIPTION:
Polycystic ovary syndrome is a disorder which is associated with insulin resistance, diabetes, obesity, and cardiovascular disease. Endothelial dysfunction, which is known to be an early marker of atherosclerosis, has also been shown to have an association with poycystic ovary syndrome. In this study the investigators aimed to investigate whether there is a relation between polycystic ovary syndrome and serum endocan levels. For this purpose the investigators designed a prospective study including two groups. The diagnosis of polycystic ovary syndrome was made in the presence of ;oligo- and/or anovulation,clinical hyperandrogenism and polycystic ovaries. Clinical hyperandrogenism was defined by the presence of hirsutism , acne, or the presence of androgenic alopecia, body mass index (BMI) was calculated as weight in kilograms divided by the square of height in meters. The two groups are compared considering their serum endocan levels,follicle stimulating hormone (FSH), luteinizing hormone (LH), Dihydroepiandesterone sulphate (DHEAS), total testesterone (TT), estradiol (E2) and thyroid stimulating hormone (TSH), fasting blood glucose, triglyceride, total cholesterol, high density lipoprotein, low density lipoprotein, and C-reactive protein (CRP) levels.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years
* Patients diagnosed with PCOS according to Rotterdam criteris (for the study group)
* Patients without PCOS and menstrual irregularities (for the control group)
* Absence of significant abnormalities on physical examination except hirsutism
* No lipid lowering, hypoglycemic, antihypertensive or hormone replacement therapy
* Normal thyroid function and prolactin level
* Absence of history or evidence of metabolic, cardiovascular, respiratory or hepatic disease

Exclusion Criteria:

* Pregnant
* Ovarian tumors
* Endocrine diseases (Cushing disease, 21-Hydroxylase enzyme deficiency, thyroid dysfunction,hyperprolactinemia,diabetes)
* Chronic diseases (renal insufficiency, cardiovascular, hepatic disease)
* Oral contraceptive use, anti-androgenic,glucocorticoid, anti-hypertansive- anti-diabetic drug use
* Smoking or alcohol use

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 84 women with PCOS and 84 healty women as control group.
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2017-01; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Serum endocan level and its relationship with Polycystic Ovary Syndrome | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ilhan B Delibas, M.D., Principal Investigator — Gaziosmanpasa University Department of Obstetrics and Gynecology; Esra Laloglu, M.D., Study Chair — Erzurum Halk Saglıgı Laboratuvarı
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)